CLINICAL TRIAL: NCT02713711
Title: Comparison of the Effectiveness of Artificial Balneotherapy, Phototherapy and Artificial Balneophototherapy in the Treatment of Psoriasis: A Randomized, Controlled Trial
Brief Title: Effectiveness of Artificial Balneotherapy, Phototherapy and Artificial Balneophototherapy in the Treatment of Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Gabriel Nasri Marzuca Nassr, PT; MSc, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUCM/1261/N822c/2014; 11/2012 (Other: Universidad Católica del Maule)
Record Dates: First submitted 2016-03-10; First posted 2016-03-21 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-01

CONDITIONS: Psoriasis
Keywords: Psoriasis; balneotherapy; phototherapy; balneophototherapy
MeSH Terms: conditions — Psoriasis | interventions — Phototherapy; Balneology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control group (No Intervention): The control group plaques did not receive any treatment.
- phototherapy group (Experimental): Twelve sessions of phototherapy (UV-B) applied on psoriatic plaques according to individual initial evaluation of Minimal Erythema Dose (MED).
  Interventions: Radiation: phototherapy
- balneotherapy (Experimental): Twelve sessions of 15 minutes of balneotherapy (warm water, 32 °C and natural sea salt, 250 g/L) applied on psoriatic plaques.
  Interventions: Procedure: balneotherapy
- balneophototherapy (Experimental): Twelve sessions of both balneotherapy and phototherapy treatments on the same conditions described above applied on psoriatic plaques.
  Interventions: Procedure: balneophototherapy

INTERVENTIONS:
Radiation: phototherapy — Twelve sessions of phototherapy (UV-B) according to individual initial evaluation of Minimal Erythema Dose (MED).
  Arms: phototherapy group
Procedure: balneotherapy — Twelve sessions of 15 minutes of balneotherapy (warm water, 32 °C and natural sea salt, 250 g/L).
  Arms: balneotherapy
Procedure: balneophototherapy — Twelve sessions of both balneotherapy and phototherapy treatments.
  Arms: balneophototherapy

SUMMARY:
The purpose of this study is to compare the effectiveness of artificial balneotherapy (AB), phototherapy (PT) and artificial balneophototherapy (BPT) in the treatment of plaque psoriasis, evaluating the plaque area, alteration of skin pigmentation, Psoriasis Area and Severity Index (PASI) score determination and quality-of-life assessment by Short Form 36 Health Survey (SF-36) and Psoriasis Disability Index (PDI) scores during the month of treatment. Methods: Experimental study, prospective, randomized, single-blind. 14 subjects participated from the city of Talca, Chile medically diagnosed with psoriasis, more than one plaque in the skin without topical treatment voluntarily. All subjects completed the study that consisted of 12 sessions.

DETAILED DESCRIPTION:
On the selected subjects, it was also performed the evaluation of Minimal Erythema Dose (MED) in order to determine an acceptable dose of UV-B light for the type of skin of each patient. Thus, the evaluations were performed according to psoriasis type, area, color and plaques severity. The formula used for the calculation was:

MED = 2×t(s)×0,75 t: minimum time for erythema occurrence.

Each psoriatic plaque was submitted to three therapeutic sessions per week, during 4 weeks, for a total of 12 sessions.

For the application of AB, the AB group plaques were immersed during 15 minutes in a 35 or 75 l hydrotherapy whirlpool (TB-T45 model and TB-T90 model respectively, Enraf Nonius Company SA, Spain) filled with a solution of warm water (32 °C) and natural sea salt (250 g/L), following the similar protocol of others authors always ensuring that the plaques not receiving this treatment were kept isolated with flexible and insulating adhesive patches (Nexcare® Factory 3M, Chile).

For the implementation of PT, the PT group plaques that would not receive radiation were covered with thick cloth towels, while the healthy skin surrounding the treated plaques were coated with liquid petroleum jelly. Both patients and attendant were protected with special lenses with filter against UV light (Oakley Jupiter, USA). UV-B radiation was applied with the UV Endolamp 474 device (Enraf Nonius Company SA, Spain), 60 cm away from the plaque and in a perpendicular position. In session 1, the MED was calculated for each subject and used as the time of UV-B exposure. On each further session, the exposure time was increased by 25%, until the limit of 5 minutes.

The BPT group plaques received both AB and PT treatments, on the same conditions described above, consecutively.

The C group plaques did not receive any treatment.

Data Collection The plaques were photographed at a distance of 20 cm with a 12 pixel Lumix digital camera (Panasonic, USA). For area quantification, the photographs were taken before session 1 and a day after session 6 and 12, and were analyzed with ImageJ software (version 1.46j; National Institute of Health, MD, USA). For color evaluation, the photographs taken before session 1 and after session 12 were analyzed with the Average color seeker software (Version 0.41; IDimager Systems Inc., Scotts Valley, CA, USA), which uses the Red-Green-Blue (RGB) coordinates system that reports the information about the red color channel, associated to erythema occurrence, in arbitrary units. Therefore, greater red color measurements for skin pigmentation may indicate increased erythema.

The psoriatic plaque severity was assessed before session 1 and one day after session 12 through PASI, which considers erythema, induration and plaque scaling, being 72 points the maximum score.

Quality of life assessment was performed using the SF-36 TM v2 health questionnaire, validated for the Chilean population10, and with the psoriasis disability index (PDI), both performed before session 1 and one day after session 12.

ELIGIBILITY:
Inclusion Criteria:

* be more than 18 years-old,
* have more than one plaque on the skin,
* medically diagnosed as plaque psoriasis over a year ago and,
* without concurrent topical treatment for Psoriasis (by own choice).

Exclusion Criteria:

* pregnancy,
* skin carcinoma,
* severe diabetes mellitus,
* uncontrolled chronic pathologies and/or severe cardiac/renal insufficiency and/or acute infections.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: psoriatic plaques
Period: Overall Study
Arm/Group | Control Group | Phototherapy Group | Balneotherapy | Balneophototherapy
Started (14 participants and 58 total psoriatic plaques divided in the 4 groups.) | 9; 14 psoriatic plaques | 6; 15 psoriatic plaques | 6; 14 psoriatic plaques | 10; 15 psoriatic plaques
Completed | 9; 14 psoriatic plaques | 6; 15 psoriatic plaques | 6; 14 psoriatic plaques | 10; 15 psoriatic plaques
Not Completed | 0; 0 psoriatic plaques | 0; 0 psoriatic plaques | 0; 0 psoriatic plaques | 0; 0 psoriatic plaques

BASELINE CHARACTERISTICS:
Population: In all the study were 14 participants with 58 total psoriatic plaques divided in 4 groups (14 in C group, 15 in AB group, 14 in PT group, and 15 in BPT group)
Units Other Than Participants: psoriatic plaques
Groups:
- All Participants: Each participant had psoriatic plaques divided into 4 groups.
  1. The control group plaques did not receive any treatment.
  2. Twelve sessions of phototherapy (UV-B) applied on psoriatic plaques according to individual initial evaluation of Minimal Erythema Dose (MED).
     - phototherapy: Twelve sessions of phototherapy (UV-B) according to individual initial evaluation of Minimal Erythema Dose (MED).
  3. Twelve sessions of 15 minutes of balneotherapy (warm water, 32 °C and natural sea salt, 250 g/L) applied on psoriatic plaques.
     - balneotherapy: Twelve sessions of 15 minutes of balneotherapy (warm water, 32 °C and natural sea salt, 250 g/L).
  4. Twelve sessions of both balneotherapy and phototherapy treatments on the same conditions described above applied on psoriatic plaques.
     * balneophototherapy: Twelve sessions of both balneotherapy and phototherapy treatments.
Arm/Group | All Participants
Number analyzed (Participants) | 14
Number analyzed (psoriatic plaques) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.85 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants] — In total were 7 male and 7 female. We divided the 58 psoriatic plaques of the 14 subjects in 4 groups (14 control group; 15 AB group; 14 PT group; 15 BPT group). A subject might have 5 psoriatic plaques, so 2 of these plaques can stay on AB group, 1 psoriatic plaque on BPT group and the last 2 on C group.
  I mean that one subject can have more than one treatment.
  Participants
    Female | 7
    Male | 7
Region of Enrollment [Number; unit: participants]
  Chile | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Psoriatic Plaque Area
Description: The plaques were photographed at a distance of 20 cm with a 12 pixel Lumix digital camera (Panasonic, USA). For area quantification, the photographs were taken before session 1 and a day after session 6 and 12, and were analyzed with ImageJ software (version 1.46j; National Institute of Health, MD, USA). A single area value was calculated per psoriatic plaque after twelve sessions (percentage of decrease).
Time Frame: Before first session (day 1), after the six session (day 12) and after the twelve session (day 26)
Population: 14 subjects (7 female and 7 male) with 58 total psoriatic plaques divided in the 4 groups
Measure: Mean (Standard Deviation); unit: percentage change
Units Other Than Participants: psoriatic plaques
Arm/Group | Control Group | Phototherapy Group | Balneotherapy | Balneophototherapy
Number analyzed (Participants) | 9 | 6 | 6 | 10
Number analyzed (psoriatic plaques) | 14 | 15 | 14 | 15
percentage change
  after session 12 | 108.22 (24.42) | 78.89 (21.04) | 84.29 (24.33) | 63.69 (21.82)
  after session 6 | 101.26 (10.81) | 84.25 (21.79) | 91.96 (18.88) | 82.09 (19.15)
Statistical Analysis 1: Comparison: Control Group; Test type: Superiority — ANOVA. Sample was calculated with power of 80% and alpha of 0.05; p = 0.3262, ANOVA; repeated measures ANOVA (Bonferroni post-test) for intragroup analysis
Statistical Analysis 2: Comparison: Phototherapy Group; Test type: Superiority — ANOVA. Sample was calculated with power of 80% and alpha of 0.05; p = 0.01, ANOVA; repeated measures ANOVA (Bonferroni post-test) for intragroup analysis
Statistical Analysis 3: Comparison: Balneotherapy; Test type: Superiority — ANOVA. Sample was calculated with power of 80% and alpha of 0.05; p = 0.0646, ANOVA; repeated measures ANOVA (Bonferroni post-test) for intragroup analysis
Statistical Analysis 4: Comparison: Balneophototherapy; Test type: Superiority — ANOVA. Sample was calculated with power of 80% and alpha of 0.05; p < 0.001, ANOVA; repeated measures ANOVA (Bonferroni post-test) for intragroup analysis
Statistical Analysis 5: Comparison: Control Group vs Phototherapy Group vs Balneotherapy vs Balneophototherapy; Test type: Superiority — Two-way ANOVA (Bonferroni post-test) for intergroup analysis; p < 0.001, ANOVA

2. Secondary Outcome: Arbitrary Units Change in Psoriatic Plaque Erythema
Description: The plaques were photographed at a distance of 20 cm with a 12 pixel Lumix digital camera (Panasonic, USA). For color evaluation, the photographs taken before session 1 and after session 12 were analyzed with the Average color seeker software (Version 0.41; IDimager Systems Inc., Scotts Valley, CA, USA), which uses the Red-Green-Blue (RGB) coordinates system that reports the information about the red color channel, associated to erythema occurrence, in arbitrary units. Therefore, greater red color measurements for skin pigmentation may indicate increased erythema. A single value was calculated per psoriatic plaque.
Time Frame: Before first session (day 1) and after the twelve session (day 26)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: arbitrary units
Units Other Than Participants: psoriatic plaques
Arm/Group | Control Group | Phototherapy Group | Balneotherapy | Balneophototherapy
Number analyzed (Participants) | 9 | 6 | 6 | 10
Number analyzed (psoriatic plaques) | 14 | 15 | 14 | 15
arbitrary units
  Before session 1 | 172.1 (28.52) | 150.2 (24.47) | 163.9 (28.13) | 159.3 (23.22)
  After session 12 | 179.4 (19.57) | 136.5 (27.50) | 154.5 (28.83) | 157.2 (30.29)
Statistical Analysis 1: Comparison: Control Group; Test type: Superiority — paired-t test (intragroup analysis); p = 0.2080, t-test, 2 sided
Statistical Analysis 2: Comparison: Phototherapy Group; Test type: Superiority — paired-t test (intragroup analysis); p = 0.0136, t-test, 2 sided
Statistical Analysis 3: Comparison: Balneotherapy; Test type: Superiority — paired-t test (intragroup analysis); p = 0.2987, t-test, 2 sided
Statistical Analysis 4: Comparison: Balneophototherapy; Test type: Superiority — paired-t test (intragroup analysis); p = 0.8347, t-test, 2 sided
Statistical Analysis 5: Comparison: Control Group vs Phototherapy Group vs Balneotherapy vs Balneophototherapy; Test type: Superiority — two-way ANOVA with Bonferroni post hoc test (intergroup analysis); p = 0.0001, ANOVA

3. Secondary Outcome: Number of Participants With Change in PASI From Baseline to Session 12
Description: The Psoriasis Area Severity Index (PASI) is an index (score determination) used to express the severity of psoriasis.
  It combines the severity (erythema, induration and desquamation) and percentage of affected area
  Instructions
  For each body section (head, arms, trunk and legs) specify:
  the percent of area of skin involved the severity of three clinical signs (erythema, induration and desquamation) on a scale from 0 to 4 (from none to maximum).
  In this study plaque severity was presented as percentage of initial value. A reduction of 75 % on plaque severity was considered effective (Puig, 2007).
Time Frame: Before first session (day 1) and after the twelve session (day 26)
Population: 14 participants
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: 14 participants with 58 psoriatic plaques divided into 4 groups.
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  PASI more than 75% | 4
  PASI more than 50% | 7
  PASI less than 50% | 3

4. Secondary Outcome: Number of Participants With Change in Quality of Life
Description: Assessment by Short Form 36 Health Survey (SF-36) score.
  The SF-36 is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. Pricing depends on the number of scores that the researcher needs to calculate.
  The eight sections are:
  vitality physical functioning bodily pain general health perceptions physical role functioning emotional role functioning social role functioning mental health
  In this study quality of life were presented as p
Time Frame: Before first session (day 1) and after the twelve session (day 26)
Population: 14 participants
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: 14 subjects with 58 psoriatic plaques divided into 4 groups.
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  Increase perception of Quality of life | 13
  Decrease perception of Quality of life | 1

5. Secondary Outcome: Number of Participants With Change in Psoriasis Disability
Description: Assessment by Psoriasis Disability Index (PDI) score.
  The Psoriasis Disability Index is calculated by summing the score of each of the 15 questions, resulting in a maximum of 45 and a minimum of 0.
  The higher the score, the more quality of life is impaired. The Psoriasis Disability Index can also be expressed as a percentage of the maximum possible score of 45.
Time Frame: Session 1 and session 12
Population: 14 participants and 58 total psoriatic plaques divided in the 4 groups
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
participants
  Improve of the autoperception of Psoriasis Disability | 13
  Maintance of the autoperception of Psoriasis Disability | 1

ADVERSE EVENTS:
Time Frame: 0 Total Number of Participants at Risk
Description: Serious and Other [Not Including Serious] Adverse Events were not collected/assessed
Arm/Group | Control Group | Phototherapy Group | Balneotherapy | Balneophototherapy
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No